CLINICAL TRIAL: NCT03737669
Title: Randomized Trial to Evaluate Mirasol Whole Blood Pathogen Reduction Technology System to Reduce Malaria and Emerging Transfusion Transmitted Infections
Brief Title: Mirasol Evaluation of Reduction in Infections Trial
Acronym: MERIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Terumo BCT (Industry); MU-JHU CARE (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00174892
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Transfusion-Transmitted Infectious Disease
Keywords: transfusion; pathogen reduction technology; Uganda; tranfusion transmitted infections; Mirasol; blood

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirasol-treated Fresh Whole Blood (Experimental): Standard Fresh Whole Blood, treated with Mirasol Pathogen Reduction Technology
  Interventions: Biological: Mirasol-treated Fresh Whole Blood
- Standard Fresh Whole Blood (Placebo Comparator): Standard-issue fresh whole blood
  Interventions: Biological: Standard Fresh Whole Blood

INTERVENTIONS:
Biological: Mirasol-treated Fresh Whole Blood — Standard issue FWB, which gave negative serological assay results for HIV, HBV, HCV, and syphilis will subsequently be treated with Mirasol PRT, then stored at 1 - 6 degrees Celsius and transfused within 21 days of collection.
  Arms: Mirasol-treated Fresh Whole Blood
Biological: Standard Fresh Whole Blood — Fresh whole blood that gave negative serological assay results for HIV, HBV, HCV, and syphilis will be stored at 1 - 6 degrees Celsius and transfused within 21 days of collection.
  Arms: Standard Fresh Whole Blood

SUMMARY:
This is a prospective, randomized, double-blind, controlled study to determine the effectiveness of Mirasol-treated fresh whole blood (FWB) versus Standard-issue FWB for preventing transmission of transfusion-transmitted infections (TTIs). The incidence of pre-defined viral, bacterial, or parasitic TTIs in previously negative participants will be assessed by changes in laboratory findings at multiple time points over the course of the clinical trial.

DETAILED DESCRIPTION:
Anemic patients from Mulago Hospital Complex who require fresh whole blood transfusion and with any of the following conditions will be considered for recruitment: cancer, general medical or surgical, obstetric hemorrhage, and/or sickle cell. Eligible patients will be randomized 1:1 to receive transfusions of Mirasol-treated FWB (n = 1,000) or standard issue FWB (n = 1,000) during the 10 week follow-up interval. The Ugandan Blood Transfusion Service collects and screens donor blood and will provide both Standard and Mirasol-treated blood for transfusion. Currently, all standard FWB is non-leukoreduced and tested by serology for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) and by rapid plasma regain (RPR) for syphilis in Uganda; any units that test positive are discarded. The intervention will treat standard FWB that has been screened for HIV, HBV, HCV, and syphilis with Mirasol PRT.

The start of study treatment (Day 0) will be defined as the initiation of the first FWB transfusion. Recipient blood collected at pre-transfusion, Day 2, Day 7, Week 4, and Week 10 will be compared with donor blood to evaluate for incidence of pre-defined TTIs: bacteria, HBV, HCV, hepatitis E virus (HEV), human herpesvirus-8 (HHV8), HIV, and malaria. Recipients will be evaluated for possible transfusion reactions at those timepoints, as well as 2 to 6 hours after the first transfusion.

The primary objective of the Uganda Mirasol Trial is to evaluate the efficacy of Mirasol-treated FWB to prevent transfusion transmission of emerging infectious diseases. The secondary objectives are to evaluate the impact of TTIs in Uganda and potential for Mirasol PRT, as well as to assess the feasibility and sustainability of implementing whole blood Mirasol pathogen reduction technology (PRT) in austere settings.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in study and patient or legally authorized representative has given written informed consent (IC)
* Hemoglobin < 7 g/dL or decision to transfusion by clinical team
* Transfusion necessary based on clinical judgment of attending physician
* Agree to return to the hospital for the follow-up visits

Exclusion Criteria:

* Presence of red cell alloantibodies
* Incompatible red cell crossmatch
* Not expected to survive for 10 weeks
* Expected to require plasma or platelets within next 10 weeks outside of the FWB provided in the trial
* Blood type AB (due to concern of limited supply)
* Weight < 30 kg (due to concern for sufficient blood draws to detect bacteria and other TTIs)
* HIV-infected
* Clinical suspicion of sepsis
* Anti-malarial treatment within 7 days prior to randomization
* Fever (central body temperature greater than 38.5°C)
* Transfusion(s) of a blood product within 1 month prior to randomization
* Acute or chronic medical disorder that, in the opinion of the investigator, would impair the ability of the patient to receive protocol treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of at least one (1) pre-defined TTI | Up to 10 weeks
  New case of any pre-defined TTIs (HIV, HBV, HCV, HEV, HHV-8, malaria, and/or bacterial infection) in a previously negative patient and matched from the blood donor, indicated by changes in laboratory findings at Day 2, Day 7, Week 4, or Week 10 after the first transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Tobian, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Mulago Hospital Complex, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kasirye R, Hume HA, Bloch EM, Lubega I, Kyeyune D, Shrestha R, Ddungu H, Musana HW, Dhabangi A, Ouma J, Eroju P, de Lange T, Tartakovsky M, White JL, Kakura C, Fowler MG, Musoke P, Nolan M, Grabowski MK, Moulton LH, Stramer SL, Whitby D, Zimmerman PA, Wabwire D, Kajja I, McCullough J, Goodrich R, Quinn TC, Cortes R, Ness PM, Tobian AAR. The Mirasol Evaluation of Reduction in Infections Trial (MERIT): study protocol for a randomized controlled clinical trial. Trials. 2022 Apr 4;23(1):257. doi: 10.1186/s13063-022-06137-8. PMID 35379302